CLINICAL TRIAL: NCT00980044
Title: Efficacy of Extended Release Tramadol for Treating Prescription Opioid Withdrawal
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Michelle Lofwall (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Michelle Lofwall, Principal Investigatory, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-0489; R01DA027068 (NIH)
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2014-12-03 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-03

CONDITIONS: Substance Withdrawal Syndrome
MeSH Terms: conditions — Substance Withdrawal Syndrome | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tramadol 200 mg then placebo (Experimental): Tramadol 200 mg daily for 1 week then placebo given for 1 week
  Interventions: Drug: Tramadol
- Placebo for two weeks (Placebo Comparator): Medication
  Interventions: Drug: Placebo
- Tramadol 600 mg then placebo (Experimental): Tramadol 600 mg daily given for 1 week given then placebo given for 1 week
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Tramadol — Oral Medication
  Other Names: Brand name example: Ultram
  Arms: Tramadol 200 mg then placebo; Tramadol 600 mg then placebo
Drug: Placebo — Oral Medication
  Other Names: Placebo is like a sugar pill
  Arms: Placebo for two weeks

SUMMARY:
Prescription opioid addiction is a growing public health problem and more pharmacologic treatments are needed because current approved medications have had limited patient acceptance (naltrexone), limited availability (methadone), and concerns about misuse and diversion (methadone and buprenorphine). Tramadol is a currently approved medication used to treat moderate-severe pain, and initial studies demonstrate that it may be useful for treatment of the uncomfortable syndrome of opioid withdrawal without producing euphoric effects. This study will determine whether two different doses of extended release tramadol can treat opioid withdrawal and whether tramadol itself produces withdrawal after it is no longer taken.

ELIGIBILITY:
Inclusion Criteria:

* Addicted to opioids

Exclusion Criteria:

* Any major medical or psychiatric disorder that would be contraindicated for participation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2009-10; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Lofwall, M.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

REFERENCES:
- [Result] Lofwall MR, Babalonis S, Nuzzo PA, Siegel A, Campbell C, Walsh SL. Efficacy of extended-release tramadol for treatment of prescription opioid withdrawal: a two-phase randomized controlled trial. Drug Alcohol Depend. 2013 Nov 1;133(1):188-97. doi: 10.1016/j.drugalcdep.2013.05.010. Epub 2013 Jun 4. PMID 23755929

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient screening. Recruitment by advertisement and word or mouth.
Pre-assignment Details: Persons screening who did not meet inclusion/ exclusion criteria were not enrolled.
  Persons who did not complete the study were not included in analyses. The study was designed as an efficacy study that a priori stated it would enroll until 12 persons in each group completed the study and analyse only completers. No serious AEs in noncompleters.
Groups:
- Tramadol 200 mg Daily: Medication: Extended release tramadol 200 mg daily given for 1 week then placebo given for 1 week
- Placebo: Placebo given for two weeks
- Tramadol 600 mg Daily: Medication: Extended release tramadol 600 mg daily given for 1 week followed by 1 week of placebo dosing.
Period: Overall Study
Arm/Group | Tramadol 200 mg Daily | Placebo | Tramadol 600 mg Daily
Started | 17 | 19 | 17
Completed | 12 | 12 | 12
Not Completed | 5 | 7 | 5
Not completed — Withdrawal by Subject | 5 | 7 | 3
Not completed — Protocol Violation | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The study was a priori defined to evaluate only completers. There were 12 completers in each of the three study arms. We retained the description of the completers because it corresponds to the primary outcomes results that are reported (and this is what was proposed a priori and approved by NIDA review).
Groups:
- Tramadol 200 mg: Medication: Extended release tramadol for 1 week and then placebo given for 1 week
- Placebo: Medication: Placebo given for two weeks
- Tramadol 600 mg: Medication: Extended release tramadol 600 mg given for 1 week and then placebo given for 1 week
- Total: Total of all reporting groups
Arm/Group | Tramadol 200 mg | Placebo | Tramadol 600 mg | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 12 | 36
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (0.9) | 32.2 (2.2) | 31.6 (1.5) | 30.1 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 5 | 14
  Male | 7 | 8 | 7 | 22
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Subjective Opioid Withdrawal Total Adjective Score
Description: range of scores is 0-84; low scores indicate no opioid withdrawal, higher scores indicating more opioid withdrawal present. T
Time Frame: Days 1-7
Population: The primary analysis was ANOVA with day and treatment arm as factors. The outcome measure described below is the mean across the days listed.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Tramadol 200 mg Daily; Tramadol 600 mg Daily: Medication: Extended release tramadol
- Placebo: Medication
Arm/Group | Tramadol 200 mg Daily | Placebo | Tramadol 600 mg Daily
Number analyzed (Participants) | 12 | 12 | 12
units on a scale | 5.8 (0.1) | 7.7 (0.1) | 6.9 (0.1)

2. Primary Outcome: Total Number of Breakthrough Withdrawal Medication Doses Taken Week 1
Description: There were four medications (acetaminophen for aches/pains, zolpidem for trouble sleeping, bismuth subsalicylate for diarrhea, and alumina/magnesia/simethicone for nausea/upset stomach) available to all volunteers in all treatment arms to help relieve any withdrawal symptoms that were not relieved by the blinded tramadol/placebo doses.
Time Frame: Days 1-7
Population: These are data from week 1 -- the 12 people who completed this week in each group. This is the analysis that was specified at the start of the study. The primary analysis was ANOVA with day and treatment arm as factors. The outcome measure described below is the mean across the days listed.
Measure: Mean (Standard Error); unit: Mean doses per day
Arm/Group | Tramadol 200 mg Then Placebo | Placebo for Two Weeks | Tramadol 600 mg Then Placebo
Number analyzed (Participants) | 12 | 12 | 12
Mean doses per day | 1.8 (0.2) | 2.5 (0.2) | 3.1 (0.3)

3. Primary Outcome: Subjective Opioid Withdrawal Adjective Total Score Week 2
Description: range of scores is 0-84; low scores indicate no opioid withdrawal, higher scores indicating more opioid withdrawal present
Time Frame: days 8-13
Population: The primary analysis was ANOVA with day and treatment arm as factors. The outcome measure described below is the mean total withdrawal score across the days listed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Tramadol 200 mg Then Placebo | Placebo for Two Weeks | Tramadol 600 mg Then Placebo
Number analyzed (Participants) | 12 | 12 | 12
units on a scale | 2.7 (0.2) | 2.9 (0.2) | 2.7 (0.1)

4. Primary Outcome: Total Number of Breakthrough Withdrawal Medication Doses Taken Week 2
Description: as for outcome 2
Time Frame: Days 8-13 (all groups now on placebo)
Population: The primary analysis was ANOVA with day and treatment arm as factors. The outcome measure described below is the mean number of doses/day across the days listed.
Measure: Mean (Standard Error); unit: mean # of doses per day
Arm/Group | Tramadol 200 mg Then Placebo | Placebo for Two Weeks | Tramadol 600 mg Then Placebo
Number analyzed (Participants) | 12 | 12 | 12
mean # of doses per day | 1.8 (0.2) | 1.6 (0.1) | 3.2 (0.2)

ADVERSE EVENTS:
Description: There were no serious adverse events for anyone enrolled (completers and non-completers). The remaining adverse events are reported from both completers and non-completers.
Groups:
- Tramadol 200 mg: Medication: Extended release tramadol 200 mg daily for one week followed by placebo for one week
- Placebo: Medication: Placebo for 2 weeks
- Tramadol 600 mg: Medication: Extended release tramadol 600 mg daily for one week followed by placebo for one week
Arm/Group | Tramadol 200 mg | Placebo | Tramadol 600 mg
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 2/17 | 1/19 | 2/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tramadol 200 mg (N=17) | Placebo (N=19) | Tramadol 600 mg (N=17)
unsteady urine flow without dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Occurred in a completer
sore throat/strep B (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Occurred in a completer
abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) — Occurred in a completer
fleeting chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Occurred in a completer
left shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Pre-existing condition -- pain due to old MVA whereby shoulder was hurt. Occurred in a non-completer.
tooth pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Cracked right front tooth prior to admission to study - now with mild pain in that tooth. Occurred in a non-completer.
flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — right sided flank pain that started 2 days prior to randomization, mild severity, occurs when twisting body. Occurred in a non-completer.
sore throat with cough (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Occurred in a non-completer.
athletes foot (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Occurred in a non-completer.

LIMITATIONS AND CAVEATS:
The study was designed to analyze only completers (12 subjects per group so the description of study participant characteristics and outcomes are from these a prior defined n=36 (12 per group) completers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No